CLINICAL TRIAL: NCT05038462
Title: Fetal Brain Care: Therapies for Brain Neurodevelopment in Fetal Growth Restriction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other); Fundació Sant Joan de Déu (Other)
Responsible Party: Principal Investigator, Elisenda Eixarch Roca, Coordinator of Fetal Neurology Unit, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Fetal Brain Care
Record Dates: First submitted 2021-08-02; First posted 2021-09-09 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Fetal Growth Retardation; Intrauterine Growth Restriction
Keywords: Fetal Growth Retardation; Fetal Growth Restriction; Intrauterine Growth Restriction; Neurodevelopment; Lactoferrin; DHA
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Lactoferrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal supplementation with Lactoferrin and DHA (Active Comparator): The intervention consists in the maternal oral administration of 1000mg of Lactoferrin and 1000mg of DHA daily
  Interventions: Dietary Supplement: Lactoferrin and DHA
- Placebo (Placebo Comparator): Product with the same physical appearance and taste as the main intervention but without therapeutic effect
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactoferrin and DHA — The intervention consists in the maternal oral administration of 1000mg of Lactoferrin and 1000mg of DHA daily
  Arms: Maternal supplementation with Lactoferrin and DHA
Other: Placebo — Product with the same physical appearance and taste as the main intervention but without therapeutic effect
  Arms: Placebo

SUMMARY:
Singleton pregnancies being diagnosed of fetal growth restriction from 24 to 32.6 weeks of gestation will be randomized to two equally sized groups: maternal oral supplementation with Lactoferrin and DHA (Docosahexaenoic acid) or placebo.

DETAILED DESCRIPTION:
Randomized controlled trial among pregnant women that have been diagnosed of fetal growth restriction. These women will be randomized in order to evaluate the impact of maternal supplementation with Lactoferrin and DHA on the neurodevelopment outcome of their babies.

Main hypothesis: a prenatal intervention based on maternal supplementation with Lactoferrin and DHA improves neurodevelopment in fetal growth restriction.

Secondary hypothesis are that a prenatal intervention based on maternal supplementation with Lactoferrin and DHA in fetal growth restriction improves fetal growth and improves perinatal morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Non-malformed fetus
* Pregnancies with fetal growth restriction
* 24-32.6 weeks of gestation

Exclusion Criteria:

* Chromosomal or structural abnormalities diagnosed during pregnancy or in the neonatal period
* Critical Doppler study suggesting the need for delivery within the next 14 days at the time of diagnosis: reverse end-diastolic velocity in the umbilical artery or ductus venosus pulsatility >95th centile
* Maternal mental or psychiatric disorders
* Maternal allergy to cow's milk protein

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bayley III scale at 24 months of age | 24 months of corrected postnatal age
  Bayley III scale is and individually administered instrument that assesses infant development across five domains, including cognitive, language and motor competencies. Parent reported questionnaires are incorporated to assess social-emotional and adaptative behaviors.

SECONDARY OUTCOMES:
Cortical development | 34 weeks of gestation
  Assessed by fetal brain magnetic resonance imaging.
Fetal brain volume | 34 weeks of gestation
  Assessed by fetal brain magnetic resonance imaging.
Corpus callosum area | Enrolment, 32 and 36 weeks of gestation
  Assessed by fetal neurosonography.
Neonatal weight | Delivery
  Birth weight
Perinatal morbidity and mortality | Perinatal period: period ranging from 32 weeks of gestation (154 days) to the end of the first 4 weeks of neonatal life (28 days)
  Development of one of the following conditions: pregnancy complications, perinatal mortality, metabolic acidosis and major neonatal morbidity.
Postnatal neurodevelopmental assessment | Between 4 and 24 months of corrected postnatal age
  Neurodevelopmental assessment using the Bayley III scale at 6 and 24 months of corrected postnatal age, as described in the primary outcome.
  A complementary neurodevelopmental assessment will be carried out in collaboration with the Speech Acquisition and Perception Groups of the University Pompeu Fabra Barcelona.
Occurrence of adverse effects | Through intervention (supplementation) completion, from enrolment to delivery
  Record of side effects that may appear. Since intervention is usually well tolerated, we do not expect major side effects.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Dexeus-Quirón, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital General del Hospitalet, L'Hospitalet de Llobregat

REFERENCES:
- See also: Related Info — http://bcnatalresearch.org/en/projects/fetalbraincare/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT05038462/Prot_SAP_002.pdf
  • Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT05038462/ICF_003.pdf